CLINICAL TRIAL: NCT04410172
Title: Prevalence of Molar Incisor Hypomineralization Among a Group Of Egyptian Children Aged From 8 to 12 Years Old in Damietta
Brief Title: Prevalence of MIH Among Group of Egyptians Children Aged From 8 to 12 in Damietta
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eman Zakaria Ali Hashem (Other)
Responsible Party: Sponsor-Investigator, Eman Zakaria Ali Hashem, B.D.S, Faculty of Dentistry, Cairo University., Cairo University
Organization: Cairo University (Other)
Other Study IDs: EMAN91
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mirror and prope — Mirror and probe will be used for each patient. Mirrors for proper visualization especially for maxillary teeth, explorers will be used to aid in tactile sensation.

SUMMARY:
Assesment of the prevalence of molar incisor hypomineralization among a group of egyptian children aged from 8 to 12 years old in Damietta governate. This study will determine the severity of molar incisor hypomineralization which will help in its managment ,also will increase the awareness pf pediatric dentists about the prevalence of molar incisor hypomineralization in Egyptian children.Also it will allow the early detection of molar incisor hypomineralization which will make the parents seek early treatment for it. Participants fromprimary schools in Damietta governate will be included in the study. Clinica examination will be carried out in the school lab or in embty class, in day light.

ELIGIBILITY:
Inclusion Criteria:

* positive subject acceptence for participation in the study.
* children aged from 8 to 12 years old.
* Eruption of at least two first permanent molars.
* Both genders.

Exclusion Criteria:

* Uncooperative child.
* Children with prthodontic appliances.
* Children with systemic diseases.
* Children suffering from any other type of enamel defect as enamel hypoplasia.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A group of Egyptian children aged from 8 to 12 years old in Damietta governate.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of molar incisor hypomineralization. | On the same day of examination
  Prevalence of molar incisor hypomineralization among a group of egyptian children aged from 8 to 12 years old. Participants will be examined in the school lab using disposable diagnostic set. Clinical examination to the four first permanent molars and the eight maxillary and mandibular incisors to detect the presence of MIH based on EAPD. To diagnose MIH, at least one affected first permanent molar is required.

REFERENCES:
- [Background] Alaluusua S. Aetiology of Molar-Incisor Hypomineralisation: A systematic review. Eur Arch Paediatr Dent. 2010 Apr;11(2):53-8. doi: 10.1007/BF03262713. PMID 20403298
- [Background] Allazzam SM, Alaki SM, El Meligy OA. Molar incisor hypomineralization, prevalence, and etiology. Int J Dent. 2014;2014:234508. doi: 10.1155/2014/234508. Epub 2014 May 8. PMID 24949012
- [Background] Biondi AM, Lopez Jordi Mdel C, Cortese SG, Alvarez L, Salveraglio I, Ortolani AM. Prevalence of molar-incisor hypomineralization (MIH) in children seeking dental care at the Schools of Dentistry of the University of Buenos Aires (Argentina) and University of la Republica (Uruguay). Acta Odontol Latinoam. 2012;25(2):224-30. PMID 23230646
- [Background] Buchgraber B, Kqiku L, Ebeleseder KA. Molar incisor hypomineralization: proportion and severity in primary public school children in Graz, Austria. Clin Oral Investig. 2018 Mar;22(2):757-762. doi: 10.1007/s00784-017-2150-y. Epub 2017 Jun 19. PMID 28631087
- [Background] Da Costa-Silva CM, Ambrosano GM, Jeremias F, De Souza JF, Mialhe FL. Increase in severity of molar-incisor hypomineralization and its relationship with the colour of enamel opacity: a prospective cohort study. Int J Paediatr Dent. 2011 Sep;21(5):333-41. doi: 10.1111/j.1365-263X.2011.01128.x. Epub 2011 Apr 6. PMID 21470321